CLINICAL TRIAL: NCT04898517
Title: Prevention of Clinically Relevant Postoperative Pancreatic Fistula in Pancreaticoduodenectomy With the Novel Technique of Connexion the Pancreatic Duct to Jejunum Stented (CONDUCTJE-ST).
Brief Title: Prevention of CR-POPF in PD With the Technique of Connexion the Pancreatic Duct to Jejunum Stented (CONDUCTJE-ST).
Acronym: CONDUCTJE-ST
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Responsible Party: Sponsor
Other Study IDs: CONDUCTJE-ST IN PD
Record Dates: First submitted 2021-05-11; First posted 2021-05-24 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Pancreas Disease; Fistula Pancreatic
Keywords: Pancreaticoduodenectomy; Postoperative pancreatic fistula
MeSH Terms: conditions — Pancreatic Diseases; Pancreatic Fistula | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pancreaticoduodenectomy with the CONDUCTJE-ST technique — The termed technique "connexion pancreatic duct to the jejunum stented" (CONDUCTJE-ST) in pancreaticoduodenectomy is a novel technique, modification of the pre-existing ones, whose effectiveness lies in the fact that it is not an anastomosis in the strict sense but rather a simple connection for restoring pancreatic juice flow from the pancreatic remnant towards the intestine.

SUMMARY:
Objective: To assess the efficacy of the "connexion pancreatic duct to jejunum stented (CONDUCTJE-ST)" technique to prevent clinically relevant postoperative pancreatic fistula (CR-POPF) after pancreaticoduodenectomy (PD).

Summary Background Data: CR-POPF remains the most determining cause of morbidity and mortality after PD. The incidence of CR-POPF (grades B and C, ISGPS) is around 20% and is a potential source of severe secondary complications that are associated with a mortality of up to 40%.

Methods: A prospective pilot study included 50 consecutive patients who underwent PD with the CONDUCTJE-ST technique, the steps of which are described, performed by the same surgical team from January 2018 to February 2020. No patient received prophylactic or therapeutic somatostatin or its analogues. The primary endpoint was the incidence of CR-POPF. Secondary endpoints were postoperative mortality and morbidity, hospital course and during the first year of follow-up.

In a prospective study we have evaluated a "novel" technique, modification of the preexisting ones, for the reconstruction of the digestive continuity of the corporocaudal remnant in the PD, termed "connexion pancreatic duct to jejunum stented (CONDUCTJE-ST)", applicable to any type of pancreatic remnant, regardless of its texture and the diameter of the main pancreatic duct. The study was planned with the objective of achieving a significant reduction in the incidence of CR-POPF, so that CONDUCTJE-ST could be considered as a surgical procedure of choice in the management of the pancreatic remnant in PD.

DETAILED DESCRIPTION:
From January 2018 to February 2020, a PD was performed with the CONDUCTJE-ST technique in 50 consecutive patients by the same surgical team, whose main surgeon has make more than 250 PD, in our Hepatobiliopancreatic Surgery and Liver Transplantation Unit. The study was carried out in accordance with the Declaration of Helsinki and was approved by the Research Ethics Committee of the Community of Aragon (CEICA), Act No. 16/2018. Patient care and study conduct complied with good clinical practices and written informed consent was obtained from each patient.

The selection of patients for surgery was decided collectively by the Multidisciplinary Committee for Tumors of the Liver, Bile ducts and Pancreas of our hospital. No patient received neoadjuvant treatment.

Technical aspects:

Patients received general anesthesia and multimodal pain therapy with an epidural catheter. All patients underwent resection with curative intent, performing PD with antrectomy and standard lymphadenectomy. Immediately after sectioning the pancreas at the level of the isthmus-body, a tissue slice is biopsied from the section margin. In the reestablishment of digestive continuity, we successively perform four reconstructions. The restoration of the flow of pancreatic juice from the corporocaudal remnant towards the intestine was carried out with the technique of "connection of the pancreatic duct to the jejunum with stent (CONDUCTJE-ST)".

Patient characteristics:

All study data were prospectively recorded. The demographic characteristics, comorbidities, clinical manifestations of the disease and intraoperative parameters were analyzed. During the intervention, the texture of the remaining pancreatic parenchyma was classified as soft or hard and the diameter of the external orifice of the main pancreatic duct was measured after transection; these data were distributed by disease pathology as confirmed by final histological assessment.

Patient outcome and follow-up. The primary endpoint of the study was the incidence of CR-POPF. No patient received prophylactic or therapeutic somatostatin or its analogues. According to the 2016 updated of the ISGPS16, POPF has been defined as any volume of fluid collected in the abdominal drainage on postoperative day 3 or from this day with an amylase level 3 times higher than the normal value serum amylase. CR-POPF has been considered when the criteria for grades B or C were met, while grade A has been replaced by the denomination of biochemical leak (16).

The volume and appearance of the fluid from the abdominal drains was recorded daily. The amylase concentration in the fluid of each of the drains was analyzed on the third and sixth postoperative days, as well as before removing the drain and on any day in which there was a substantial increase in volume or change in the appearance of the fluid. The drains were removed when three requirements were met: amylase levels in the drainage fluid less than 8 twice the plasma level (normal 28-100 U / L), volume <25 ml / day, and clear appearance of the fluid.

The secondary endpoints of the study were: 1) postoperative mortality, defined as that which occurred within thirty days of the operation or during the same hospital admission; 2) postoperative complications related to the surgical technique: delayed gastric emptying (DGE), digestive and intra-abdominal hemorrhage, intra-abdominal abscesses, surgical wound infection, biliary fistula and gastrointestinal fistula; 3) days of stay in the Intensive Care Unit (ICU) and hospital, reoperations, and readmissions. The DGE and postoperative bleeding were defined according to the ISGPS29,30. The severity of complications was classified using the Clavien-Dindo system31; a severe complication was defined as grade IIIa or higher; 5) during the first year after PD: a) the incidence of exocrine pancreatic insufficiency (EPI), evaluated by the presence of steatorrhea, need for pancreatic enzyme supplements and fecal elastase determination; b) incidence of new-onset diabetes mellitus (NODM), assessed by blood glucose, glycated hemoglobin A1c and need for insulin or oral antidiabetics; c) overall survival and by pathologies and, in the case of malignant processes, disease-free survival, at 3, 6, 9 and 12 months after PD.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years
* informed surgical and anesthetic consents
* scheduled surgical intervention
* intention to carry out PD with the CONDUCTJE-ST technique

Exclusion Criteria:

* emergency PD
* performing another pancreatic resection technique other than PD
* associated resection of another viscus
* metastasis or locally advanced unresectable tumor detected during surgery.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in whom a pancreaticoduodenectomy (PD) is to be performed due to carcinoma of the pancreas head, distal common bile duct, biliopancreatic confluent and duodenum. Also in neuroendocrine tumors and pancreatic cystic neoplasms such as intraductal papillary mucinous neoplasia and mucinous cystadenoma, and in some forms of chronic pancreatitis.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of clinically relevant postoperative pancreatic fistula after pancreaticoduodenectomy | From surgery up to 30 days after pancreaticoduodenectomy
  According to the 2016 updated of the ISGPS16, POPF has been defined as any volume of fluid collected in the abdominal drainage on postoperative day 3 or from this day with an amylase level 3 times higher than the normal value serum amylase. CR-POPF has been considered when the criteria for grades B or C were met, while grade A has been replaced by the denomination of biochemical leak. The volume and appearance of the fluid from the abdominal drains was recorded daily. The amylase concentration in the fluid of each of the drains was analyzed on the third and sixth postoperative days, as well as before removing the drain and on any day in which there was a substantial increase in volume or change in the appearance of the fluid.

SECONDARY OUTCOMES:
Postoperative mortality | From surgery to 30 days after pancreaticoduodenectomy
  Defined as that which occurred within thirty days of the operation
Delayed gastric emptying (DGE) | From surgery up to 30 days after pancreaticoduodenectomy
  Defined according to the ISGPS
Postoperative hemorrhage | From surgery up to 30 days after pancreaticoduodenectomy
  Defined according to the ISGPS
Severity of postoperative complications | From surgery up to 30 days after pancreaticoduodenectomy
  Classified using the Clavien-Dindo system31; a severe complication was defined as grade IIIa or higher
Incidence of exocrine pancreatic insufficiency | One year after pancreaticoduodenectomy.
  Evaluated by the presence of steatorrhea, need for pancreatic enzyme supplements and fecal elastase determination
Incidence of new-onset diabetes mellitus | One year after pancreaticoduodenectomy.
  Assessed by blood glucose, glycated hemoglobin A1c and need for insulin or oral antidiabetic

CONTACTS AND LOCATIONS:
Overall Officials: Francisco A. García-Gil, MD, Principal Investigator — Instituto de Investigación Sanitaria Aragón
Locations (1):
- University Clinic Hospital Lozano Blesa, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No